CLINICAL TRIAL: NCT01621945
Title: Phase 3, Vaccinal Activity Assessment of MenBVac Against Neisseria Meningitidis B:14,P1.7,16 Strain in Child
Brief Title: Evaluation of Immune Response Against the Strain of Neisseria Meningitidis B: 14, P1-7, 16 in Patients Having to be Vaccinated MenBVac® (Extension EFFIVAC)
Acronym: Exten Effivac
Status: Completed | Type: Observational
Sponsor: University Hospital, Rouen (Other)
Collaborators: Direction Générale de la Santé, France (Other); Institut Pasteur (Industry)
Responsible Party: Sponsor
Other Study IDs: 2011/198/HP
Record Dates: First submitted 2012-03-26; First posted 2012-06-18 (Estimated); Last update posted 2014-09-08 (Estimated); Status verified 2014-09

CONDITIONS: Neisseria Meningitidis
Keywords: Neisseria meningitidis B:14, P1-7, 16; Serum bactericidal activity; OMV vaccine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Bras A: children, born between the 06/04/2004 and the 17/04/2008, living around Neufchatel en Bray, before the fourth dose of MenBVac
  Interventions: Biological: MenBvac

INTERVENTIONS:
Biological: MenBvac — Blood test

SUMMARY:
The main objective of the study is to estimate the proportion of children, born between the 06/04/2004 and the 17/004/2008, living around Neufchatel en Bray, vaccinated by MenBVac, with a serum bactericidal activity against B:14,P1-7,16 clone related to a protection (>= 4), before the fourth dose of MenBvac and after: 6 weeks and one year after the fourth dose.

ELIGIBILITY:
Inclusion Criteria:

* children born between 06/04/2004 and 17/04/2008, living in Neufchatel en Bray,and Having participated to the first study,
* children who Have to be Vaccinated MenBVac® for the four times,
* parental authority(ies)assent.

Exclusion Criteria:

* no parental authority(ies)assent,
* no blood sample,
* impossibility of fourth vaccination,
* children yet vaccinated or non eligible for vaccination.

Ages: 4 Years to 8 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Children aged 4 to 8 years old and living in neufchatel en bray area
Sampling Method: Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2012-04; Primary Completion 2013-04 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Vaccine Immunity | after the fourth dose of MenbVac
  Assessment of vaccine Immunity with measure of percentage of children who have hSBA title >= 4 six weeks after the fourth dose of vaccine

CONTACTS AND LOCATIONS:
Locations (1):
- Maison Du Département, Neufchâtel-en-Bray, France